CLINICAL TRIAL: NCT07060963
Title: Evaluation of the Effect of Pender's Health Promotion Theory Based Diabetes Self-Management Program on Healthy Living Behaviors in Pregnant Women Diagnosed With Gestational Diabetes Mellitus
Brief Title: Evaluation of Healthy Lifestyle Behaviors in Pregnant Women Diagnosed With Gestational Diabetes Mellitus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Esra Altun, NURSE, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-84892257-300-292369
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Self-Efficacy for Decision Making; Apgar Score; Behavior Change; Maternal and Neonatal Outcomes; Models, Theoretical
Keywords: Gestational diabetes; nursing; motivational interviewing,; diabetes management; health promotion theory
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interviewing within the context of a health promotion-based diabetes mellitüs (Active Comparator): The group that received the diabetes self-management program based on the Pender's health promotion model
  Interventions: Behavioral: Motivational interviews within the context of a health promotion-based diabetes self-management program
- Routine maintenance standard (No Intervention): The group that did not receive the diabetes self-management program based on Pender's health promotion model

INTERVENTIONS:
Behavioral: Motivational interviews within the context of a health promotion-based diabetes self-management program — The researcher provided counseling services to pregnant women to provide Diabetes Self-Management Group training based on Pender's Health Promotion Model. A group was formed consisting of at least 10 people. The training was completed face-to-face and practically, in 1 day (160 minutes), in 4 sessions, each session being 40 minutes. Motivational interviews were conducted by the researcher within the scope of the health promotion-based diabetes self-management program. A second motivational interview was planned according to the determined need and the interviews were provided. Each interview lasted approximately 40 minutes. In order to ensure continuity for the pregnant women who obtained positive behavioral outcomes, reinforcement was provided by telephone interviews and the counseling process was completed.
  Arms: Motivational interviewing within the context of a health promotion-based diabetes mellitüs

SUMMARY:
The aim was to evaluate the effect of a nursing education intervention based on Pender's SGM on gestational diabetes management and healthy lifestyle behaviors for pregnant women diagnosed with gestational diabetes. The main questions it aims to answer are:

1. Is there a difference between the total mean scores of the Healthy Lifestyle Behaviors Scale of the pregnant women in the intervention and control groups?
2. Is there a difference between the total mean scores of the Self-Efficacy in Gestational Diabetes Scale of the pregnant women in the intervention and control groups?
3. Is there a difference between the total mean scores of the Health Belief Model Scale in Diabetic Patients of the pregnant women in the intervention and control groups?
4. Is there a difference between the total mean scores of the Multidimensional Perceived Social Support Scale of the pregnant women in the intervention and control groups?
5. Is there a difference between the development of maternal complications (at least one complication) of the pregnant women in the intervention and control groups?
6. Is there a difference in the development of fetal complications (at least one complication) between the pregnant women in the intervention and control groups?

DETAILED DESCRIPTION:
It was conducted in the Department of Obstetrics and Gynecology (GHD) of the Cebeci Application and Research Hospital (AÜTFCH) of Ankara University Faculty of Medicine. This study was conducted with pregnant women who were diagnosed with OGTT test at 24-28 weeks of pregnancy and applied to the AÜTFCH GHD pregnancy clinic.

The study was conducted in two stages: the first stage was the preparation of research materials and determination of study groups, and the second stage was the implementation of the diabetes self-management program based on the Penderin health promotion model.

In the first stage of the study, women diagnosed with gestational diabetes mellitus (GDM) who constituted the intervention and control groups were divided into groups using the simple randomization method. Patients diagnosed according to the oral glucose tolerance test (OGTT) results are started to be followed up in the perinatology clinic. Pregnant women are routinely referred to a dietician in the perinatology clinic. In order to prevent bias, support was received from a dietician independent of the study to create an intervention and control group. Randomization was used to prevent distribution bias. Patients who applied to the dietician were grouped according to their application days. Patients formed the intervention group on the 1st, 3rd and 5th days of the first week, while the control group formed the 2nd and 4th days. The control group formed the 1st, 3rd and 5th days of the second week, while the intervention group formed the 2nd and 4th days. The education groups were divided into groups of at least 10 people by taking into account their gestational weeks. The second phase of the study included the application of the Diabetes Self-Management Program Based on Pender's Health Promotion Model to the pregnant women in the intervention group. Face-to-face interviews were conducted with pregnant women in the intervention group who were diagnosed with gestational diabetes and were between 24-28 weeks of pregnancy. Pregnant women who agreed to participate in the study were informed about how the study would proceed and their written consent was obtained. The pregnant women in the intervention group were asked to fill out the personal information form and the pre-test (Health Belief Model Scale in Diabetic Patients (DHSMÖ), Gestational Diabetes Self-Efficacy Scale (GDSES), Healthy Lifestyle Behaviors-II Scale (HLBS-II), Multidimensional Perceived Social Support Scale (MSPSS)]. Their contact information was obtained to facilitate the follow-up process of the pregnant women and to organize the training program. The researcher determined the day and time of the training according to the availability of the pregnant women to provide the Diabetes Self-Management Group training based on Pender's Health Promotion Model. The group was formed with at least 10 people. The first group completed the training with 16 people, the second group with 11 people, and the third group with 14 people. The training was completed face-to-face and practically, in 4 sessions of 1 day (160 minutes), each session being 40 minutes. In order to support the training program, the "Training for Patients with Gestational Diabetes Booklet", and to ensure follow-up and continuity, the "Lifestyle Behavior Change Follow-up Booklet" was given to the pregnant women and its use was explained. They were asked to bring the follow-up booklet to each interview, and the researcher determined the motivational interview topics according to the DHSMÖ sub-dimension scores and the booklet. In line with the interviews, motivational interviews were conducted within the scope of the health development-based diabetes self-management program by the researcher who has a certificate in diabetes life coaching, holistic medicine eating and drinking disorders and motivational interview. The first motivational interview was conducted between the 32nd and 34th weeks of pregnancy for each pregnant woman in the intervention group according to their DHSMÖ and HLBS-II scale sub-dimension scores. Before each interview, the pregnant women were called by phone to remind them of the interview. A follow-up file was created for each pregnant woman. The follow-up file includes OGTT test results, lifestyle behavior change booklet, DHSMÖ sub-dimension scores, motivational interview schedules, pre-test and post-test forms.

A second motivational interview was planned between the 32nd and 36th weeks of pregnancy according to the determined need situation and the pregnant women were asked to repeat the relevant DHSMÖ sub-dimension. were provided. Each interview lasted approximately 40 minutes. During the study, group dynamics were maintained by having the pregnant women post walking videos and photos of their meals. In order to ensure continuity for the pregnant women who achieved positive behavioral outcomes, reinforcement was provided by phone calls and the counseling process was completed.

ELIGIBILITY:
Inclusion Criteria:

* Able to communicate in Turkish,
* Not having conditions that would create communication problems (mental, visual, hearing impairment),
* Graduated from at least secondary school,
* Having a singleton pregnancy between the 24th and 28th weeks of pregnancy,
* Not having been diagnosed with GDM in a previous pregnancy,
* Not having been diagnosed with a risky pregnancy (adolescent pregnancy, preeclampsia, eclampsia, hypertension),
* Not having a health problem that would prevent exercise (heart disease, respiratory diseases, risk of abortion, orthopedic problems),
* Not having to follow a special diet program (Celiac disease, kidney disease, heart disease).
* Not having a psychiatric diagnosis (psychosomatic disorders),
* Having an endocrine disease known to affect blood glucose levels (hyperthyroidism, hypothyroidism).

Exclusion Criteria:

* Wanting to leave at any stage of the study,
* Not participating in the program at least once after joining the study (Signature chart follow-up, detection of non-continuation of daily follow-up),
* Being diagnosed with a risky pregnancy at any stage of the study (preeclampsia, eclampsia, premature membrane rupture, systemic disease)
* Incompletely filling in the data collection forms applied during the program.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 68 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Health Belief Model Scale in Diabetic Patients | It is applied between the 24th-28th weeks of pregnancy and the 38th-40th weeks of pregnancy
  Both medical and non-medical methods are used in the treatment management of gestational diabetes mellitus. The scale used in the study was developed to evaluate the health beliefs and attitudes of diabetic patients and to examine their health behaviors. The scale consists of 33 items. According to the results of the factor analysis, it was determined that the scale consists of five sub-dimensions.- Perceived susceptibility: - Perceived seriousness: - Perceived benefits: - Perceived barriers: - It evaluates recommended activities related to health. The subscale mean score is obtained by summing the items for each subscale and dividing by the number of items in the relevant subscale. A score of four or more indicates high (positive) health beliefs, while a score of less than four indicates low (negative) health beliefs.The lowest score for the entire scale is 33 and the highest score is 165.
Self-Efficacy Scale in Gestational Diabetes | It is applied between the 24th-28th weeks of pregnancy and the 38th-40th weeks of pregnancy
  The self-efficacy scale for gestational diabetes was developed based on four dimensions: "Diet-weight management," "Complication precautions," "Adherence to nutrition education," and "Medical treatment practices." In the overall assessment of the scale, based on the overall mean score obtained from the item mean scores of all subscales, those with scores below the mean were considered to have low self-efficacy, while those with scores above the mean were considered to have high self-efficacy. The lowest score for the entire scale was 23, and the highest was 115.
Healthy Lifestyle Behaviors Scale - II | It is applied between the 24th-28th weeks of pregnancy and the 38th-40th weeks of pregnancy
  The scale consists of 52 items and six factors. Subscales;
  * Health responsibility
  * Physical activity
  * Nutrition
  * Spiritual development
  * Interpersonal relationships
  * Stress management. The lowest score for the entire scale is 52, the highest score is 208. An increase in the score obtained from the scale indicates a better level of healthy lifestyle behaviors
Multidimensional Perceived Social Support Scale | It is applied between the 24th-28th weeks of pregnancy and the 38th-40th weeks of pregnancy
  The scale consists of 12 items. Each of the scales consists of three subscales, each consisting of four items, related to the source of support. These subscales are family, friends, and a special person. The subscale score is obtained by adding the scores of the four items in each subscale, and the total score of the scale is the total score. The lowest score to be obtained from the subscales is 4, the highest score is 28, and the lowest score to be obtained from the total scale is 12, the highest is 84. A high score indicates that perceived social support is high. A score of 42 and above from the scale, which can be scored between 12 (worst) and 84 (best), indicates that there is a positive situation regarding social support.

SECONDARY OUTCOMES:
Postpartum Follow-up Form | It will be evaluated within 24-48 hours after birth.
  The birth outcomes for the mother and baby will be examined within the first 24-48 hours after birth and postpartum. The planned hospital stay for the study is at least 24 hours for normal birth and 48 hours for cesarean section. Before the patient is discharged, maternal and fetal postpartum outcomes (delivery method, mother's innatal and postpartum blood serum glucose levels, baby's birth weight, baby's APGAR scores, baby's blood serum glucose levels, complications for the mother and newborn) will be evaluated from the patient files.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt Üniversitesi, Sağlık Bilimleri Fakültesi, Ankara, Çubuk, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-09-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT07060963/ICF_000.pdf